CLINICAL TRIAL: NCT06108219
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Miricorilant in Adult Patients With Nonalcoholic Steatohepatitis/Metabolic Dysfunction-Associated Steatohepatitis (MONARCH)
Brief Title: A Phase 2b, Study Evaluating Miricorilant in Adult Patients With Nonalcoholic Steatohepatitis/Metabolic Dysfunction-Associated Steatohepatitis (MONARCH)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CORT118335-862
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Metabolic Dysfunction-associated Steatohepatitis (MASH)
Keywords: Nonalcoholic Steatohepatitis (NASH); Nonalcoholic Fatty Liver Disease (NAFLD); Metabolic dysfunction-Associated Steatohepatitis (MASH); Metabolic dysfunction-Associated Steatosis Liver Disease (MASLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — CORT118335

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Experimental (Cohort A) (Experimental): Patients who meet the entry criteria for study CORT118335-862 (Cohort A) will be enrolled to receive 100 mg of miricorilant, twice a week for 48 weeks.
  Interventions: Drug: Miricorilant (Cohort A)
- Placebo (Cohort A) (Placebo Comparator): Patients who meet the entry criteria for study CORT118335-862 (Cohort A) will be enrolled to receive a matching placebo twice a week for 48 weeks.
  Interventions: Drug: Placebo (Cohort A)
- Placebo (Cohort B) (Placebo Comparator): Patients who meet the entry criteria for study CORT118335-862 (Cohort B) will be enrolled to receive a matching placebo twice a week for 24 weeks.
  Interventions: Drug: Placebo (Cohort B)
- Experimental (Cohort B) (Experimental): Patients who meet the entry criteria for study CORT118335-862 (Cohort B) will be enrolled to receive 100 mg of miricorilant, twice a week for 6 weeks. Dose will be escalated to 200 mg of miricorilant, twice a week for 18 weeks.
  Interventions: Drug: Miricorilant (Cohort B)

INTERVENTIONS:
Drug: Miricorilant (Cohort A) — Miricorilant 100 mg for oral dosing
  Other Names: CORT118335
  Arms: Experimental (Cohort A)
Drug: Placebo (Cohort A) — Matching placebo for oral dosing for 48 Weeks
  Arms: Placebo (Cohort A)
Drug: Miricorilant (Cohort B) — Miricorilant 100 mg for oral dosing Miricorilant 200 mg for oral dosing
  Other Names: CORT118335
  Arms: Experimental (Cohort B)
Drug: Placebo (Cohort B) — Matching placebo for oral dosing for 24 Weeks
  Arms: Placebo (Cohort B)

SUMMARY:
A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Miricorilant in Adult Patients with Nonalcoholic Steatohepatitis (MONARCH)

DETAILED DESCRIPTION:
Approximately 75 patients who are eligible for participation in the study will be randomized on Day 1 in a 2:1 ratio to 100 mg miricorilant or placebo twice weekly, for 48 weeks of treatment (Cohort A).

Approximately 90 patients who are eligible for participation in the study will be randomized on Day 1 in a 2:1 ratio to 100 mg miricorilant twice a week for 6 weeks of treatment, followed by a dose escalation to 200 mg miricorilant or placebo twice weekly for an additional 18 weeks which resulting in a total treatment duration of 24 weeks, or to placebo for 24 weeks. (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Histological diagnosis of NASH/MASH with NAS ≥ 4 (≥ 1 point in each subcomponent of steatosis, inflammation, and ballooning) and NASH-CRN fibrosis score of 2 or 3 based on the consensus method of histological assessment. A historical liver biopsy within 6 months of Screening with reading confirmed during the Screening period by a consensus panel is acceptable.
* Cohort B: Have a liver biopsy result that does not meet with the criteria for inclusion in Cohort A and is consistent with one of the following based on the consensus method of histological assessment:

  * NAS ≥ 3 with ≥1 point in each subcomponent of steatosis, inflammation, and ballooning, and a NASH-CRN fibrosis score of F1 or
  * NAS ≥ 2 with ≥1 point in subcomponent of steatosis and ≥ 1 point in subcomponent of ballooning or inflammation and a NASH-CRN fibrosis score of F2 or 3
* AST > 17 U/L for women and AST > 20 U/L for men.
* FibroScan® liver stiffness measurement ≥ 8 kPa and CAP ≥ 280 dB/m.
* MRI-PDFF with ≥ 8% steatosis
* Presence of at least 1 of the following metabolic syndromes that increase the risk of NASH/MASH:

  1. Diagnosis of type 2 diabetes OR
  2. Presence of 2 or more components of metabolic syndrome:

  i. Fasting blood glucose ≥ 100 mg/dL (5.6 mmol/L) or treatment for elevated blood glucose ii. Systolic blood pressure ≥ 130mmHg, diastolic blood pressure ≥ 85mmHg, or treatment for hypertension iii. Serum triglycerides ≥ 150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides iv. Serum high-density lipoprotein (HDL) cholesterol < 40 mg/dL (1 mmol/L) in men and < 50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL v. Overweight or obese (body mass index [BMI] ≥ 25 kg/m2 [BMI ≥ 23 kg/m2 in Asians]), or increased waist circumference ≥ 102 cm (40 in) in men and ≥ 88 cm (35 in) in women (male ≥ 90 cm [35.4 in]; women ≥ 80 cm [31.5 in] in
* Other inclusion criteria may apply

Exclusion Criteria:

* Have participated in another clinical trial within the last 3 months of Screening where the patient received active treatment for NASH/MASH.
* Have participated in a clinical trial for any other indication within the last 3 months or 5 half-lives of the treatment, whichever is longer.
* Are pregnant or lactating women
* Have a BMI < 18 kg/m2 or > 45 kg/m2.• Have had liver transplantation or plan to have liver transplantation during the study
* Have type 1 diabetes or poorly controlled type 2 diabetes.
* Are pregnant or lactating women
* Have a BMI < 18 kg/m2 or > 45 kg/m2
* Have had successful weight-loss surgery within 2 years prior to Screening or are planning weight-loss surgery during the study.
* Have a >5% weight change within 3 months prior to Screening.
* Have significant alcohol consumption of more than 20 g per day for women and 30 g per day for men within 1 year prior to screening or score of ≥8 on AUDIT questionnaire
* Have any other chronic liver disease
* History of cirrhosis or evidence of cirrhosis by clinical, imaging, or liver biopsy evaluation
* Have hepatic decompensation
* Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent relative change from Baseline in liver-fat content assessed by MRI-PDFF (Cohort A and Cohort B) | Week 24

SECONDARY OUTCOMES:
Change in liver stiffness and Controlled Attenuation Parameter (CAP) by FibroScan. (Cohort A and Cohort B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in absolute body weight (Cohort A and B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in lipids - total cholesterol, HDL, LDL, VLDL, TG, serum free fatty acids, apolipoproteins (Cohort A and Cohort B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) (Cohort A and Cohort B at Week 6 and 24, Cohort A at Week 48) | Week 6, 24 and 48
Change in ELF, Pro-C3 and other markers of liver fibrosis (Cohort A and B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in HbA1c (Cohort A and B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in HOMA-IR (Cohort A and B at Week 24, Cohort A at Week 48) | Week 24 and 48
Change in plasma glucose (Cohort A and B at Week 24, Cohort A at Week 48) | Week 24 and 48
Percent relative change from Baseline in liver-fat content by MRI-PDFF (Cohort A and B at Week 6 and 24, Cohort A at Week 48) | Week 6 and 24, Week 48
Absolute change from Baseline in liver-fat content by MRI-PDFF (Cohort A and B at Week 6 and 24, Cohort A at Week 48) | Week 6, 24, Week 48
Resolution of steatohepatitis (defined as a ballooning grade of 0 and a lobular inflammation grade of ≤ 1) and no worsening of liver fibrosis at Week 48 assessed by biopsy (Cohort A). | Week 48
Proportion of patients with at least 2 points reduction from Baseline in the NAS (NAFLD activity score) without worsening of liver fibrosis at Week 48 assessed by biopsy, with at least a 1-point reduction in ballooning or inflammation (Cohort A). | Week 48
Improvement in liver fibrosis stage by at least 1-point (NASH CRN fibrosis score) from Baseline and no worsening of steatohepatitis at Week 48 assessed by biopsy (Cohort A). | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (77):
- United States (48):
  - Site #207, Chandler, Arizona
  - Site #209, Tucson, Arizona
  - Site #378, Huntington Park, California
  - Site #439, Lancaster, California
  - Site #469, Long Beach, California
  - Site #373, Los Angeles, California
  - Site #214, Panorama City, California
  - Site #233, Santa Ana, California
  - Site #452, Boca Raton, Florida
  - Site # 101, Gainesville, Florida
  - Site #465, Hallandale, Florida
  - Site #430, Hialeah Gardens, Florida
  - Site #458, Lakewood Rch, Florida
  - Site #475, Largo, Florida
  - Site #438, Miami Lakes, Florida
  - Site #460, Viera, Florida
  - Site #453, Houma, Louisiana
  - Site #451, Marrero, Louisiana
  - Site #061, Metairie, Louisiana
  - Site #440, Rockville, Maryland
  - Site #442, Saint Paul, Minnesota
  - Site #228, Kansas City, Missouri
  - Site #455, Jackson, New Jersey
  - Site #445, East Syracuse, New York
  - Site #454, New York, New York
  - Site #464, Morehead City, North Carolina
  - Site #447, Beavercreek, Ohio
  - Site #470, Columbus, Ohio
  - Site #448, Dayton, Ohio
  - Site #437, Westlake, Ohio
  - Site #461, Cordova, Tennessee
  - Site # 546, Arlington, Texas
  - Site #545, Austin, Texas
  - Site #211, Austin, Texas
  - Site #432, Brownsville, Texas
  - Site #370, Dallas, Texas
  - Site #213, Edinburg, Texas
  - Site #215, Edinburg, Texas
  - Site #431, Georgetown, Texas
  - Site # 066, Houston, Texas
  - Site #305, Houston, Texas
  - Site #459, Katy, Texas
  - Site #433, San Antonio, Texas
  - Site #212, San Antonio, Texas
  - Site #434, Waco, Texas
  - Site #441, West Jordan, Utah
  - Site #463, Manassas, Virginia
  - Site #226, Seattle, Washington
- India (28):
  - Site #506, Guwahati, Assam
  - Site #492, Ahmedabad, Gujarat
  - Site #513, Rajkot, Gujarat
  - Site #490, Surat, Gujarat
  - Site #514, Surat, Gujarat
  - Site #502, Vadodara, Gujarat
  - Site # 494, Rohtak, Haryana
  - Site #511, Mysore, Karnataka
  - Site #507, Thiruvananthapuram, Kerala
  - Site #512, Mumbai, Maharashtra
  - Site #509, Mumbai, Maharashtra
  - Site #500, Nagpur, Maharashtra
  - Site #496, Pune, Maharashtra
  - Site #495, Ludhiana, Punjab
  - Site #489, Jaipur, Rajasthan
  - Site # 485, Jaipur, Rajasthan
  - Site #508, Madurai, Tamil Nadu
  - Site #486, Hyderabad, Telangana
  - Site #549, Lucknow, Uttar Pradesh
  - Site #488, Varanasi, Uttar Pradesh
  - Site #503, Varanasi, Uttar Pradesh
  - Site #504, Dehradun, Uttarakhand
  - Site #487, Kolkata, West Bengal
  - Site #493, Kolkata, West Bengal
  - Site #491, Kolkata, West Bengal
  - Site #482, New Delhi
  - Site #510, New Delhi
  - Site #501, New Delhi
- Site #457, San Juan, Puerto Rico